CLINICAL TRIAL: NCT04269525
Title: Clinical Research Regarding the Availability and Safety of UC-MSCs Treatment for Serious Pneumonia and Critical Pneumonia Caused by the 2019-nCOV Infection
Brief Title: Umbilical Cord(UC)-Derived Mesenchymal Stem Cells(MSCs) Treatment for the 2019-novel Coronavirus(nCOV) Pneumonia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZhiYong Peng (Other)
Collaborators: Tuohua Biological Technology Co. Ltd (Unknown)
Responsible Party: Sponsor-Investigator, ZhiYong Peng, professor, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020002
Record Dates: First submitted 2020-02-07; First posted 2020-02-13 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Pneumonia, Viral; Pneumonia, Ventilator-Associated
Keywords: 2019-nCOV infection; UC-MSCs Treatment
MeSH Terms: conditions — Pneumonia, Viral; Pneumonia, Ventilator-Associated; COVID-19

STUDY DESIGN:
Intervention Model Description: reaching the criteria of pneumonia according to Diagnosis and Clinical Management of Pneumonia caused by 2019-nCoV Infection(Trial Version 4)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pneumonia (Experimental): According to Diagnosis and Clinical Management of Pneumonia caused by 2019-nCoV Infection(Trial Version 4), patients enrolled will be divided to serious pneumonia group or critical pneumonia group. All subjects will receive UC-MSCs 3.3 * 107 cell number / 50ml / bag, 3 bags each time. And UC-MSCs will be infused intravenously on the 1st, 3rd, 5th, and 7th days after enrollment, 1 time each day. The efficacy and safety of the treatment, patients' adverse reactions will be monitored.
  Interventions: Biological: UC-MSCs

INTERVENTIONS:
Biological: UC-MSCs — After enrollment, each subject will receive UC-MSCs infusion intravenously on day 1, day 3, day 5, and day 7.

SUMMARY:
Serious Pneumonia and Critical Pneumonia caused by the 2019-nCOV infection greatly threats patients' life, UC-MSCs treatment has been proved to play a role in curing multiple diseases. And this study is conducted to find out whether or not it will function in 2019-nCOV infection Pneumonia.

DETAILED DESCRIPTION:
Serious Pneumonia and Critical Pneumonia caused by the 2019-nCOV infection greatly threats patients' life, UC-MSCs treatment has been proved to play a role in curing multiple diseases. And this study is conducted to find out whether or not it will function in 2019-nCOV infection Pneumonia. And we are going to get the permission of the enrolled patients. Besides the present clinical treatment, UC-MSCs treatment will be applied to those fulfilling the enrollment. After a period of UC-MSCs treatment, the analysis of UC-MSCs treatment will be completed from related aspects.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old ,no gender restriction
* According to Diagnosis and Clinical Management of Pneumonia caused by 2019-nCoV infection(Trial Version 6), patients are diagnosed with severe or critical 2019-nCoV pneumonia
* Women of childbearing age should have a negative blood pregnancy test before the start of dosing and agree to take effective contraceptive measures during the trial until the last follow-up (28 days)
* Previous detection of Nucleotide or antibody of 2019-nCoV pneumonia was positive
* Voluntarily participate in this clinical study and sign a written informed consent. If the patient cannot obtain informed consent, he can authorize his legal representative.

Exclusion Criteria:

* Liver SOFA score of more than 3 points;
* HIV positive
* Highly allergic constitution or history of severe allergies;
* Pregnant and lactating women;
* Patients with malignant tumors;
* Patients with previous history of pulmonary embolism;
* Participating in clinical trials of other drugs within 3 months before enrollment.
* be thought by researchers to be inappropriate to participate in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Oxygenation index | on the day 14 after enrollment
  partial arterial oxygen pressure (PaO2) / oxygen concentration (FiO2)

SECONDARY OUTCOMES:
28 day mortality | on the day 28 after enrollment
  whether the patient survives
Hospital stay | up to 6 months
  days of the patients in hospital
2019-nCoV antibody test | on the day 7,14,28 after enrollment
  whether or not the 2019-nCoV antibody is positive
2019-nCoV nucleic acid test | on the day 7,14,28 after enrollment
  whether or not the 2019-nCoV nucleic acid test is positive
Improvement of lung imaging examinations | on the day 7,14,28 after enrollment
  whether lung imaging examinations show the improvement of the pneumonia
White blood cell count | on the day 7,14,28 after enrollment
  counts of white blood cell in a litre of blood
Lymphocyte count | on the day 7,14,28 after enrollment
  counts of lymphocyte in a litre (L) of blood
Procalcitonin | on the day 7,14,28 after enrollment
  procalcitonin in microgram(ug)/L
interleukin(IL)-2 | on the day 7,14,28 after enrollment
  IL-2 in picogram(pg)/millilitre(mL)
IL-4 | on the day 7,14,28 after enrollment
  IL-4 in pg/mL
IL-6 | on the day 7,14,28 after enrollment
  IL-6 in pg/mL
IL-10 | on the day 7,14,28 after enrollment
  IL-10 in pg/mL
tumor necrosis factor(TNF)-α | on the day 7,14,28 after enrollment
  TNF-α in nanogram(ng)/L
γ-interferon(IFN) | on the day 7,14,28 after enrollment
  γ-IFN in a thousand unit (KU)/L
C-reactive protein(CRP) | on the day 7,14,28 after enrollment
  CRP in microgram（μg）/L
CD4+ T-Lymphocytopenia | on the day 7,14,28 after enrollment
  counts of CD4+ T-Lymphocytopenia in litre
CD8+ T-Lymphocytopenia | on the day 7,14,28 after enrollment
  counts of CD8+ T-Lymphocytopenia in a litre
natural killer cell(NK) | on the day 7,14,28 after enrollment
  counts of NK in a litre

CONTACTS AND LOCATIONS:
Overall Officials: XingHuan Wang, professor, Study Chair — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No